CLINICAL TRIAL: NCT07125183
Title: A Phase II Study on Efficacy and Tolerability of Weekly Doxorubicin in Elderly Patients With Advanced or Metastatic Leiomyosarcoma of Soft Tissue
Brief Title: Study on Efficacy and Tolerability of Weekly Doxorubicin in Elderly Patients With Advanced or Metastatic Leiomyosarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0118.cc; NCI-2025-05219 (Other: CTRP)
Record Dates: First submitted 2025-07-18; First posted 2025-08-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma
Keywords: Metastatic Sarcoma; Advanced Sarcoma; leiomyosarcoma; doxorubicin; geriatric
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma | interventions — Doxorubicin; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doxorubicin (Experimental): Doxorubicin will be administered on days 1 and 8 every 21 days for a maximum of 8 cycles (Cycles 1-8) with appropriate premedications and pegfilgrastim growth factor support. Doxorubicin will be administered as a bolus infusion on day 1 and day 8 with dexrazoxane cardioprotection. Patients must have central line access for this protocol, including pheresis or trifusion catheter, PICC line, or port.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin is an antibiotic derived from the Streptomyces peucetius bacterium. It has widespread use as a chemotherapeutic agent since the 1960s. Doxorubicin is part of the anthracycline group of chemotherapeutic agents. Doxorubicin may be used to treat soft tissue and bone sarcomas and cancers of the breast, ovary, bladder, and thyroid. It is also used to treat acute lymphoblastic leukemia, acute myeloblastic leukemia, Hodgkin lymphoma, and small cell lung cancer.
  Other Names: Lipodox; Lipodox 50; Doxil

SUMMARY:
The overall goal of this Phase 2 study is to determine the efficacy of a lower dose weekly schedule of doxorubicin in patients with unresectable leiomyosarcomas aged 65-100 years old. While doxorubicin is the standard of care therapy for sarcomas not removable by surgery, older or more frail patients may struggle to tolerate side effects of the treatment including immune cell suppression. Previous studies have suggested that similar anti-tumor activity can be obtained using a lower dose, weekly administration schedule of doxorubicin. In this study, the investigators will determine progression-free survival rate at 12 weeks, with secondary endpoints including quality of life and adverse events in this population. Importantly, doxorubicin can also induce immune stimulatory effects when administered at lower doses, based on animal data. Thus, correlative samples including blood and tumor biopsies will also explore the effects of immune cells and foreignness of the tumor prior to and during treatment in study patients.

DETAILED DESCRIPTION:
The study is an open-label, single-arm, investigator-initiated Phase 2 trial enrolling up to 30 patients to obtain 20 evaluable patients with advanced/metastatic leiomyosarcomas. The study will utilize a time-to-event Bayesian optimal Phase 2 design. The design includes one interim futility look after 10 patients are evaluable for progression-free survival rate at 12 weeks. The outcomes will be compared to historical PFS 12 week rate calculated as the mean from two large randomized Phase 3 studies. The treatment will be deemed promising if the number of patients who are stable at 12 weeks is 65%. Early stopping rules for toxicity are included in addition to futility.

The primary endpoint of the study is the PFS rate at 12 weeks with secondary endpoints including PFS at 6 months, response rate by RECIST 1.1, duration of response, overall survival, adverse events, and quality of life scores. Correlative studies will include analysis of serial blood samples and baseline and on-treatment tumor biopsies for immune markers including analysis of tumor-infiltrating lymphocytes, tumor immune pathways, analysis of circulating immune cells, and plasma cytokines.

Following informed consent and screening, patients will receive doxorubicin 25 mg/m2 administered by bolus with dexrazoxane pre-treatment on days 1 and 8 every 21 days for up to 8 cycles. Patients will receive pegfilgrastim growth factor on day 9. Scans for response imaging will be obtained every 6 weeks during the treatment portion of the study, then every 12 weeks after completing treatment up to 1 year. Patients will have routine safety labs, assessment of adverse events, quality of life questionnaires with treatment visits, and echocardiogram to assess for cardiac toxicity will be performed at cycle 4 of doxorubicin and at the completion of study therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be male or female aged 65-100 years at the time of signing informed consent.
4. Have a histological diagnosis of advanced or metastatic soft tissue leiomyosarcoma (LMS) (by local pathology review), not curable by surgery, for which treatment with weekly doxorubicin is deemed appropriate by the investigator.
5. Have measurable or non-measurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors. Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is documented, or a biopsy is obtained to confirm persistence at least 90 days following completion of radiotherapy.
6. Have received 0 to 4 prior systemic therapies for metastatic sarcoma and NO prior anthracyclines. Re-treatment with the same drug or regimen after interruption (i.e. chemotherapy holiday) is not considered a new line of treatment, and those patients are eligible.
7. Adequate organ function
8. ECOG performance status of 0, 1 or 2.
9. Patients must consent and be willing to undergo tumor core needle biopsies at two time points: 1. Baseline, 2. Cycle 2 Day 1 (+/- 7 days); a third biopsy for off-study/progression is optional but advised. At least one tumor site must be amenable to biopsy in the judgment of the interventional radiologist and/or inverstigator.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Prior history of vasectomy does NOT replace requirement for contraceptive use.
11. Female subjects will be post-menopausal as evidenced by cessation of menses for a minimum of 2 years. Prior hysterectomy or bilateral oophorectomy is also permissible.
12. Subjects must either possess or undergo placement of central venous catheter, including pheresis or trifusion catheter, PICC line, or port.

Exclusion Criteria:

1. Prior therapy with anthracycline.
2. Hypersensitivity to doxorubicin or any excipients.
3. Patients may not be receiving any other investigational agents (within 28 days prior to Cycle 1, Day 1).
4. Patient has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 21 days prior to Cycle 1, Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 21 days earlier. Subjects with ≤ Grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study.

   Note: If a subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Additional known malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
6. Patients with underlying immune deficiency, chronic infections including hepatitis, and known history of HIV or tuberculosis (TB).
7. Patients with underlying hematologic issues including bleeding diathesis, such as known previous GI bleeding requiring intervention within the past 6 months. Newly diagnosed pulmonary emboli or deep venous thrombosis must be clinically stable on anticoagulation regimen for ≥ 2 weeks as of Cycle 1 Day 1.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease. Subjects with previously treated brain metastases may participate provided they are stable based on the following: 1) MRI brain obtained during screening evaluations shows no radiographic evidence of progression or new lesions, 2) any neurologic symptoms have returned to baseline. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability. Patients without a known history of brain metastases do not require screening brain MRI prior to study enrollment.
9. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
10. Any uncontrolled, intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
11. Prolonged QTc interval on Screening EKG >475 ms.
12. Left Ventricular Ejection Fraction <50% by 2D ECHO or MUGA scan at Screening.
13. Any serious medical or psychiatric illness/condition including substance use disorders likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment, including NYHA Class II or greater heart disease.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of treatment measured by Progression Free Survival (PFS) rate at 12 weeks | 12 weeks
  weekly doxorubicin chemotherapy in anthracycline-naïve patients measured through PFS at 12 weeks by RECIST 1.1

SECONDARY OUTCOMES:
Progression Free Survival rate at 6 months | 6 month
  Rate of patients that are progression-free at the 6 month timepoint by RECIST 1.1
Quality of Life (QoL) by EORTC-QLQ-30 | 6 months
  Patients will complete questionnaires to assess clinical benefit. The assessment will be based on a scale of strongly agree to strongly disagree.
Quality of Life by QLQ-ELD14 | 6 months
  Patients will complete questionnaires to assess clinical benefit. The assessment will be based on a scale of strongly agree to strongly disagree.
Response rate measured by RECIST 1.1 | 18 months
  Response rate by RECIST 1.1. Scans will be obtained every 6 weeks while on study therapy.
Duration of Response | 18 months
  Time that patients achieve a partial or complete response until progression by RECIST 1.1.
Overall Survival | 18 months
  Length of time from study enrollment to death by any cause.
Proportion of Doxorubicin Doses administered. | 6 months
  Evaluable patients will receive at least one dose of doxorubicin. We will determine the proportion of doses administered according to the study protocol, that are not omitted due to toxicity.
Toxicity Assessed by Adverse Events | 6 months
  Adverse events will be assessed using CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Breelyn Wilky, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University Of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No